CLINICAL TRIAL: NCT01732211
Title: A PHASE 2 RANDOMIZED, DOUBLE BLIND, PLACEBO CONTROLLED, PARALLEL GROUP, 20-WEEK SAFETY, TOLERABILITY, AND EFFICACY STUDY OF PD 0360324 IN ADULT SUBJECTS WITH CHRONIC PULMONARY SARCOIDOSIS
Brief Title: A Phase 2, Safety, Tolerability, and Efficacy Study of PD 0360324 in Chronic Pulmonary Sarcoidosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: A6261009
Record Dates: First submitted 2012-11-19; First posted 2012-11-22 (Estimated); Results first posted 2020-01-06 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2019-12

CONDITIONS: Pulmonary Sarcoidosis
Keywords: Phase 2; Randomized; Double Blind; Placebo Controlled; Parallel; 20 Week Safety; Tolerability; and Efficacy Study
MeSH Terms: conditions — Sarcoidosis, Pulmonary | interventions — Saline Solution; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PD 0360324 (Experimental)
  Interventions: Biological: PD 0360324
- Placebo (Placebo Comparator)
  Interventions: Other: Normal Saline for injection

INTERVENTIONS:
Biological: PD 0360324 — 100 mg Q2W or 150 mg Q2W via intravenous infusion based on protocol determined dose escalation/de-escalation criteria; 12 weeks Active Therapy;
  Arms: PD 0360324
Other: Normal Saline for injection — normal saline Q2W via intravenous infusion for 12 weeks
  Arms: Placebo

SUMMARY:
The study proposes to evaluate the safety, tolerability, and efficacy of PD 0360324 in subjects with chronic pulmonary sarcoidosis inadequately treated with standard of care therapies.

DETAILED DESCRIPTION:
The trial was terminated prematurely on Mar 24, 2014 due to a business decision. The decision to terminate the trial was not based on any clinical safety or efficacy concerns.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of biopsy-proved chronic pulmonary sarcoidosis either Stage 2 or Stage 3 for at least 1 year;
* Forced Vital Capacity (FVC) lung assessment of >40% and < or = to 80% predicted normal values at screening;
* age 21-75 years of age;
* treatment with a stable (longer than 4 weeks) regimen of corticosteroids (between 10 and 30 mg of prednisone) for at least 3 months prior to Screening; (other anti-inflammatory drugs may be permitted as defined by the study protocol)

Exclusion Criteria:

* History of any other pulmonary (lung) disease than sarcoidosis (ex, asthma requiring maintenance treatment, chronic obstructive pulmonary disease (COPD));
* Pulmonary hypertension, significant lung fibrosis, any chronic infection (eg, TB, HIV);
* treatment with other biologic anti-inflammatory/immuno-modulatory drugs;
* active smokers;
* class 3 or 4 congestive heart failure;
* cancer, or history of cancer within past 5 years;
* history of ischemic heart disease, heart attack, stroke, any heart muscle disease;
* liver disease;
* history of alcohol or drug abuse

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-03-15 (Actual); Primary Completion 2013-09-23 (Actual); Study Completion 2013-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- United States (5):
  - Mount Sinai School Of Medicine/Mount Sinai Medical Center, New York, New York
  - Medical Arts Building, Cincinnati, Ohio
  - The Barrett Cancer Center at UC Health, Cincinnati, Ohio
  - University Hospital, Cincinnati, Ohio
  - Iinterstitial Lung Disease & Sarcoidosis Clinic, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6261009&StudyName=A%20Phase%202%2C%20Safety%2C%20Tolerability%2C%20and%20Efficacy%20Study%20of%20PD%200360324%20in%20Chronic%20Pulmonary%20Sarcoidosis

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In Part A, approximately 22 subjects were to be enrolled to receive PD 0360324 100 mg once every 2 weeks (Q2W)/150 mg Q2W. In Part B, approximately 66 subjects were planned to be enrolled to receive PD 0360324 (either 100 or 150 mg Q2W defined in Part A) B.
Groups:
- PD 0360324 100 mg Q2W / 150 mg Q2W: PD-0360324 100 milligram (mg) was administered as intravenous infusion on Day 1 of every 2 weeks for Week 0 and Week 2. PD-0360324 150 mg was administered as intravenous infusion on Day 1 of every 2 weeks for Weeks 4, 6, 8, 10, and 12.
Period: Overall Study
Arm/Group | PD 0360324 100 mg Q2W / 150 mg Q2W
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | PD 0360324 100 mg Q2W / 150 mg Q2W
Number analyzed (Participants) | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (NA) — Standard deviation cannot be calculated for a sample size of 1.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (Absolute) in % Predicted Forced Vital Capacity (FVC) Compared to Placebo at Week 16
Description: The percent predicted FVC was calculated by observed FVC/predicted FVC * 100. The predicted FVC values was calculated according to age, height, race and gender. FVC is the volume of air which can be forcibly exhaled from the lungs after taking the deepest breath possible.
Time Frame: Baseline, Week 16
Population: No subjects were analyzed due to early termination of the study and the small enrollment number.
Arm/Group | PD 0360324 100 mg Q2W / 150 mg Q2W
Number analyzed (Participants) | 0

2. Secondary Outcome: Change From Baseline in Chest X-ray Global Assessment Score (5-point )
Description: Digital copies of Chest x-rays performed during the study were graded according to a 5 point Likert scale: 1 = markedly worsened; 2 = worsened; 3 = unchanged; 4 = improved; and 5 = markedly improved. Baseline will be defined as the last available x-ray prior to first dose.
Time Frame: Baseline, Week 16
Population: No subjects were analyzed due to early termination of the study and the small enrollment number.
Arm/Group | PD 0360324 100 mg Q2W / 150 mg Q2W
Number analyzed (Participants) | 0

3. Secondary Outcome: Change From Baseline in FVC (Absolute ) Compared to Placebo at Weeks 2,4,8,12, 14, and 20
Description: FVC is the volume of air which can be forcibly exhaled from the lungs after taking the deepest breath possible. Trough FVC was obtained from spirometry, performed before study treatment administration.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 14, and 20
Population: No subjects were analyzed due to early termination of the study and the small enrollment number.
Arm/Group | PD 0360324 100 mg Q2W / 150 mg Q2W
Number analyzed (Participants) | 0

4. Secondary Outcome: Change From Baseline Absolute in FVC (% Predicted) Compared to Placebo at Weeks 2,4,8,12,14, and 20
Description: as for outcome 1
Time Frame: Baseline, Weeks 2, 4, 8, 12, 14, and 20
Population: No subjects were analyzed due to early termination of the study and the small enrollment number.
Arm/Group | PD 0360324 100 mg Q2W / 150 mg Q2W
Number analyzed (Participants) | 0

5. Secondary Outcome: Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1) at Weeks 2,4,8,12,14, 16 and 20
Description: FEV1 is the maximal volume of air exhaled in the first second of a forced expiration from a position of full inspiration. Trough FEV1 was obtained from spirometry, performed before study treatment administration.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 14, 16, and 20
Population: No subjects were analyzed due to early termination of the study and the small enrollment number.
Arm/Group | PD 0360324 100 mg Q2W / 150 mg Q2W
Number analyzed (Participants) | 0

6. Secondary Outcome: Change From Baseline in % Predicted FEV1 at Weeks 2,4,8,12,14, 16 and 20
Description: The percent predicted FEV1 was calculated by observed FEV1/predicted FEV1 * 100. The predicted FEV1 values was calculated according to age, height, race and gender. FEV1 is the maximal volume of air exhaled in the first second of a forced expiration from a position of full inspiration.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 14, 16, and 20
Population: No subjects were analyzed due to early termination of the study and the small enrollment number.
Arm/Group | PD 0360324 100 mg Q2W / 150 mg Q2W
Number analyzed (Participants) | 0

7. Secondary Outcome: Change From Baseline in Ratio of FEV1/FVC at Weeks 2,4,8,12,14, 16 and 20
Description: FEV1 is the maximal volume of air exhaled in the first second of a forced expiration from a position of full inspiration. Trough FEV1 was obtained from spirometry, performed before study treatment administration. FVC is the volume of air which can be forcibly exhaled from the lungs after taking the deepest breath possible. Trough FVC was obtained from spirometry, performed before study treatment administration.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 14, 16, and 20
Population: No subjects were analyzed due to early termination of the study and the small enrollment number.
Arm/Group | PD 0360324 100 mg Q2W / 150 mg Q2W
Number analyzed (Participants) | 0

8. Secondary Outcome: Estimated Treatment Effect Over Placebo in FVC Averaged Over 16 Weeks
Description: FVC is the volume of air which can be forcibly exhaled from the lungs after taking the deepest breath possible. Through FVC was obtained from spirometry, performed before study treatment administration.
Time Frame: Baseline, Weeks 0, 2, 4, 8, 12, 14, 16
Population: No subjects were analyzed due to early termination of the study and the small enrollment number.
Arm/Group | PD 0360324 100 mg Q2W / 150 mg Q2W
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | PD 0360324 100 mg Q2W / 150 mg Q2W
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PD 0360324 100 mg Q2W / 150 mg Q2W (N=1)
Eye swelling (Eye disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1

LIMITATIONS AND CAVEATS:
Due to early termination of the study and the small enrollment number, analysis of primary and secondary pharmacodynamic endpoints could not be performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.